CLINICAL TRIAL: NCT06097650
Title: Cold Snare Polypectomy Versus Hot Snare Polypectomy for the Resection of Small Pedunculated Colorectal Polyps: a Multicentre Randomised Controlled Trial
Brief Title: Cold Snare Polypectomy Versus Hot Snare Polypectomy for Resection of Small Pedunculated Polyps
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Collaborators: Ninghai Second Hospital (Unknown); The People's Hospital of Yuyao City (Unknown); The Third People's Hospital Health Care Group of Cixi (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-140A-YJ01
Record Dates: First submitted 2023-10-18; First posted 2023-10-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Pedunculated Colorectal Polyps; Haemorrhage
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cold snare polypectomy (Experimental): cold snare polypectomy for resection of small pedunculated colorectal polyps
  Interventions: Other: cold snare polypectomy
- hot snare polypectomy (Active Comparator): hot snare polypectomy for resection of small pedunculated colorectal polyps
  Interventions: Other: hot snare polypectomy

INTERVENTIONS:
Other: cold snare polypectomy — Histological analyses suggest that cold snare polypectomy causes less damage to blood vessels in the submucosal layers, which results in a reduced incidence of hemorrhage
  Arms: cold snare polypectomy
Other: hot snare polypectomy — According to current clinical guidelines, hot snare polypectomy is the recommended standard technique for the resection of pedunculated colorectal polyps.
  Arms: hot snare polypectomy

SUMMARY:
Endoscopic resection of pedunculated polyps mainly focuses on how to prevent bleeding, and also needs to pay attention to the convenience of resection and the integrity of resection, which means that different endoscopic resection strategies should be adopted for pedunculated polyps with different stalk sizes. Small pedunculated polyps with heads smaller than 20mm and stalks less than or equal to 5mm are defined as having a relatively small risk of bleeding. Preliminary studies in recent years suggest that the use of cold snare polypectomy for small pedunculated polyps may also be a safe resection strategy. However, for small pedunculated polyps, ASGE and ESGE guidelines currently recommend hot snare polypectomy in the middle and lower pedicles (evidence level medium). Therefore, the provision of high-quality clinical evidence related to cold resection techniques in the resection strategy of small pedunculated polyps may provide a basis for revision of guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients undergoing endoscopic resection of small pedicled polyps in the First Affiliated Hospital of Ningbo University, The Third People's Hospital Health Care Group of Cixi, Ninghai Second Hospital and Renmin Hospital of Yuyao City from October 2023 to August 2026; 2. Patients who voluntarily agreed to participate in this study and signed informed consent.

Exclusion Criteria:

* 1. Persons under 18 years of age 2. Persons unwilling or unable to provide informed consent 3. Treatment or radiotherapy for malignant diseases, severe chronic heart or lung diseases, coronary or cerebrovascular events requiring hospitalization within the last 3 months 4.polyps with endoscopic features suspicious for carcinoma 5. Abdominal symptoms such as severe abdominal pain, abdominal distension, and nausea 6.Patients with inadequate intestinal preparation 7. Patients with lifelong anticoagulant therapy or severe bleeding diseases, patients who have recently taken anticoagulant drugs or antiplatelet drugs (within 1 week) 8.Pregnant or lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
delayed hemorrhage | 2 days, 2 weeks and 4 weeks
  Any symptoms of gastrointestinal bleeding (e. g. hematochezia) occurred within 30 days after polypectomy and were classified as mild or severe according on the severity of the bleeding

SECONDARY OUTCOMES:
Prevalence of immediate bleeding | 1 Minutes
  Immediate bleeding was defined as an intraoperative bleeding immediately after Immediate bleeding staging: If there is no bleeding, fill in 'none'; Level 1, spontaneous hemostasis within 60 seconds; Level 2, continuous small bleeding for more than 60 seconds; Level 3, continuous bleeding for more than 60 seconds requires endoscopic treatment; Level 4, arterial spray

OTHER OUTCOMES:
Immediate perforation rate | Immediate
  perforation

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang, China